CLINICAL TRIAL: NCT06686238
Title: Acute Effects of a Hypoxia-hyperoxia Exposure Session on Sedentary Older Adults on Heart Rate Variability, Blood Pressure, and Oxygen Saturation, a Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Acute Effects of Intermittent Hypoxia-Hyperoxia in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 015
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Older Adults; Cardiovascular Health; Blood Pressure; Sedentary
Keywords: hypoxic exposure; older adults; heart rate variability
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxic-Hyperoxic group (Experimental): The EG (Experimental Group) will undergo a single session of IHHE (Intermittent Hypoxia-Hyperoxia Exposure) session using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany). They will breathe air with an oxygen concentration (FiO2) ranging from 10-14% for 5 minutes, followed by 3 minutes of rest in hyperoxia (FiO2 30-40%), for a total of 6 cycles. During the hypoxic phase, oxygen saturation will be maintained between 85-92%, while during the hyperoxic phase, it will be kept above 95%. This process is regulated by the device's AI.
  Participants will be asked to sit and breath normally in each exposure.
  An attendance checklist will be used to monitor compliance with the intervention
  Interventions: Device: MITOVIT® Hypoxic Training System
- Sham Hypoxic-Hyperoxic Group (Sham Comparator): The Sham Group (SG) will follow a single session protocol of 5 cycles of 6 minutes per session with an FiO2 of 21% using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany).
  Participants will be asked to sit and breath normally in each exposure.
  An attendance checklist will be used to monitor compliance with the placebo intervention.
  Interventions: Device: Sham MITOVIT® Hypoxic Training System

INTERVENTIONS:
Device: MITOVIT® Hypoxic Training System — The EG (Experimental Group) will undergo a single session of IHHE (Intermittent Hypoxia-Hyperoxia Exposure) session using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany). They will breathe air with an oxygen concentration (FiO2) ranging from 10-14% for 5 minutes, followed by 3 minutes of rest in hyperoxia (FiO2 30-40%), for a total of 6 cycles. During the hypoxic phase, oxygen saturation will be maintained between 85-92%, while during the hyperoxic phase, it will be kept above 95%. This process is regulated by the device's AI. Participants will be asked to sit and breath normally in each exposure. An attendance checklist will be used to monitor compliance with the intervention
  Other Names: Hypoxic-Hyperoxic Exposure
  Arms: Hypoxic-Hyperoxic group
Device: Sham MITOVIT® Hypoxic Training System — The Sham Group (SG) will follow a single session protocol of 5 cycles of 6 minutes per session with an FiO2 of 21% using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany). Participants will be asked to sit and breath normally in each exposure. An attendance checklist will be used to monitor compliance with the placebo intervention.
  Other Names: Sham Hypoxic-Hyperoxic Exposure
  Arms: Sham Hypoxic-Hyperoxic Group

SUMMARY:
The supply of oxygen is essential for energy production, recovery from efforts, and human life. Intermittent Hypoxia-Hyperoxia Exposure (IHHE) is a novel technique in which the subject is exposed to a respiratory environment with reduced oxygen fraction, controlled through a specific software, using a facial mask and a hypoxic generation device. The objective of this study is to determine if there is a relationship between intermittent hypoxia-hyperoxia exposure and cardiorespiratory condition, blood pressure, and arterial oxygen saturation.

According to our hypothesis, acute IHHE in elderly adults may influence cardiorespiratory condition, blood pressure, and arterial oxygen saturation.

The study will be conducted as a randomized clinical trial. The subjects will be divided into two groups: the experimental group will undergo an IHHE session, breathing air with an oxygen concentration (FiO2) ranging from 10-14% for 1-5 minutes, with 1-3 minutes of rest in hyperoxia (FiO2 30-40%) for a total of 4-8 cycles, based on their acute response to hypoxia. The placebo group will undergo a 5-cycle protocol with an FiO2 of 21%.

ELIGIBILITY:
Inclusion Criteria:

* Being over 60 years old.
* Having no previous experience in hypoxic training.
* Engaging in less than 150 minutes of physical activity per week.

Exclusion Criteria:

* Having any pathology that prevents the subject from being independent in terms of walking and functionality.
* Subjects with impaired cognitive abilities.
* Subjects with pulmonary hypertension, decompensated heart or respiratory disease.
* To have or have had cancer

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-12-05 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-26 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | Immediately before intervention and immediately after intervention
  The analysis of Heart Rate Variability will be conducted using a heart rate monitor. Cardiac electrical signals will be monitored with a band placed on the chest for 5 minutes with the subject in supine position on a stretcher, in a quiet environment, soft light, and a comfortable temperature. Subjects are instructed not to speak or make voluntary movements during this analysis.

SECONDARY OUTCOMES:
Blood pressure | Immediately before intervention and immediately after intervention
  Both systolic and diastolic blood pressure will be assesed using a standard digital sphygmomanometer (Omron HEM-705CP, Omron Healthcare, Inc, Lake Forest, IL)
Arterial oxygen saturation | Immediately before intervention and immediately after intervention
  Arterial oxygen saturation will be assessed using a device Nonin® 3230 (Nonin Medical, Inc. Plymouth, MN, EEUU)

CONTACTS AND LOCATIONS:
Locations (1):
- Residencial Montes de Toledo, Manzaneque, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Yes